CLINICAL TRIAL: NCT06725173
Title: Genetic Associations of Ocular Cancers
Brief Title: Detailed Phenotypic and Genotype Study to Correlate RB1 Mutations Relating to Primary Ocular Tumors and Secondary Extra-ocular Metastasis.
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Debarshi Mustafi, Assistant Professor: School of Medicine, Ophthalmology, University of Washington
Other Study IDs: STUDY00021737; K08EY033789 (NIH)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Retinoblastoma Bilateral; Retinoblastoma Unilateral; Retinoblastoma, Extraocular; Retinoblastoma, Recurrent; Retinoblastoma
Keywords: retinoblastoma; parent-of-origin
MeSH Terms: conditions — Retinoblastoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extract DNA from saliva or blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with presumed germline retinoblastoma due to RB1 mutation
  Interventions: Genetic: Targeted Long-read sequencing

INTERVENTIONS:
Genetic: Targeted Long-read sequencing — All patient's will undergo targeted long-read sequencing to resolve genomic and epigenomic signatures of the RB1 gene
  Other Names: Long-read sequencing

SUMMARY:
The goal of this observational study is undertake a detailed phenotypic and genotypic study of patients with ocular and secondary cancers due to mutations in the RB1 gene. Our research sequencing approach will allow advanced insight to for further detailed genotypic understanding of parent-of-origin for valuable insight into the genotype-phenotype relationship of this cancer syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with molecularly proven retinoblastoma due to RB1 or a typical clinical retinoblastoma phenotype with genetic screening pending.
* Able to give consent/parent or guardian able to give consent.

Exclusion Criteria:

* Patients unable or unwilling to undertake consent or clinical testing.
* Patients unwilling to donate a saliva or blood sample in order to establish the genetic cause of their condition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with presumed or genetically confirmed retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Epigenomic and genomic profiling of the RB1 gene | 5 years
  Methylation signatures and genomic variant information to determine phase of the pathogenic variants in RB1 to specific differentially methylated signals in RB1

CONTACTS AND LOCATIONS:
Overall Officials: Debarshi Mustafi, MD PhD, Principal Investigator — University of Washington; Andrew W Stacey, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stacey AW, Nakamichi K, Huey J, Stevens J, Waligorski N, Crotty EE, Van Gelder RN, Mustafi D. Prognostic importance of direct assignment of parent of origin via long-read genome and epigenome sequencing in retinoblastoma. JCI Insight. 2024 Dec 26;10(4):e188216. doi: 10.1172/jci.insight.188216. PMID 39724000
- [Background] Nakamichi K, Stacey A, Mustafi D. Targeted long-read sequencing allows for rapid identification of pathogenic disease-causing variants in retinoblastoma. Ophthalmic Genet. 2022 Dec;43(6):762-770. doi: 10.1080/13816810.2022.2141797. Epub 2022 Nov 3. PMID 36325802
- See also: Related Info — https://www.mustafilab.org/